CLINICAL TRIAL: NCT06655597
Title: A 12-week Randomized, Controlled, Clinical Trial Evaluating the Efficacy of a Dietary Supplement Powder Formula (Daily Ultimate Essentials) in an Adult Population.
Brief Title: Efficacy of a Dietary Supplement Powder Formula (Daily Ultimate Essentials) in an Adult Population.
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Prenetics Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR20240501
Record Dates: First submitted 2024-10-19; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Dietary Assessment
Keywords: Dietary Supplement; Healthy Adults

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reds Powder (Experimental): Reds Powder
  Interventions: Dietary Supplement: REDS Powder
- Standard (No Intervention): Usual Diet

INTERVENTIONS:
Dietary Supplement: REDS Powder — Dietary supplement powder
  Arms: Reds Powder

SUMMARY:
Healthy Adult subjects

DETAILED DESCRIPTION:
The study will be a prospective randomized, controlled clinical study. There will be interventional treatment for a total of 12 weeks. The subjects will attend two appointments in the clinic throughout the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 30 kg/m2
* Low, moderate, and high activity (self-identified) *
* Self-identify as having fatigue, and abdominal issues (bloating, constipation etc.) *
* Participants will be able to read, understand and sign an informed consent form (includes HIPAA and States requirements) and sign a photo release form.
* Participants are willing and able to follow all study directions, attend study visits as scheduled and must be willing to accept the restrictions of the study including but not limited to:
* Willing to refrain from introducing any new diets or dietary supplements for the duration of the study

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-02-14 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Body Morphology | 12 weeks
  Subjects assessed through weight and height which will be combined to determine BMI and abdominal and thigh circumference and images before and after

SECONDARY OUTCOMES:
Safety and Tolerability | 12 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Energy | 12 weeks
  Assessed by subjective questionnaire
Changes in Micronutrient blood levels | 12 weeks
  Assessed through laboratory assays of vitamins and minerals in the blood

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco Research Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
deidentified data will be shared with data analysis team
Supporting Information: SAP, Analytic Code
Time Frame: end of the trial - 2/2025 through end of analysis 5-25
Access Criteria: Data team will access data through encrypted password protected central server and it will be all raw data and subject numbers and blinding code